CLINICAL TRIAL: NCT04937361
Title: Monitoring of MDRO Dynamics and Resistance Mechanisms in a University Hospital Network
Acronym: R-Net
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Collaborators: University Hospital of Berlin (Other); University Hospital of Cologne (Other); University Hospital Freiburg (Other); University of Giessen (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Nadja Käding, Dr. med., University of Luebeck
Other Study IDs: DZIF TTU 08.824
Record Dates: First submitted 2021-06-10; First posted 2021-06-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: MDRO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Bacterial strains isolated from rectal swabs, blood cultures and samples derived thereof (such as purified DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rectal swab — collection of rectal swabs

SUMMARY:
Survey on the prevalence of MDRO to monitor the import of MDRO from the community. Rectal swabs will be taken and cultivated. Survey on community-onset and nosocomial bloodstream infections will be documented and strains will be isolated. For each BSI a clinical data set will be obtained (e.g. patient age, gender, date of hospitalization, antibiotic therapy). Genetic analysis of MDRO from the prevalence and BSI study. In a subset of patients the microbiome-resistome interactome will be analysed in more detail. Furthermore, the impact of infection control measures due to the Covid-19 pandemic on nosocomial BSI will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* informed consent
* inpatient

Exclusion Criteria:

* less than 18 years old
* Not capable of giving informed consent
* outpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the prevalence, adult patients admitted to the hosptial within the last 3 days.
  For BSI surveillance, adult inpatients with at least one blood culture positive for any of the target organisms: Staphylococcus aureus, Enterococcus spp., Escherichia coli, Enterobacter spp., Klebsiella spp., Acinetobacter baumannii, Pseudomonas aeruginosa.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
monitoring of MDRO prevalence | at hospital admission
  obtain a better understanding for the emergence of resistance within the microenvironment under selective pressure
monitoring of blood stream infections | during hospitalization, up to 4 weeks
  obtain a better understanding for the emergence of resistance within the microenvironment under selective pressure
integrate novel techniques for microbiome-resistome interaction analysis | through study completion, after 4 years
  obtain a better understanding for the emergence of resistance within the microenvironment under selective pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Infektiologie und Mikrobiologie, Lübeck, Germany